CLINICAL TRIAL: NCT01278355
Title: The Feasibility of Integrating Ear Acupuncture for Pain in Patients Being Transported Via the Aeromedical Evacuation System From Ramstein Air Base to Andrews AFB, Maryland USA: An Observational Study
Brief Title: Assessing the Feasibility of Integrating Ear Acupuncture Into the Aeromedical Evacuation System From RAB to AAFB
Status: Completed | Type: Observational
Sponsor: Samueli Institute for Information Biology (Other)
Responsible Party: Sponsor
Other Study IDs: C.2010.041dt
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2012-12

CONDITIONS: Musculoskeletal Pain
Keywords: pain; acupuncture
MeSH Terms: conditions — Musculoskeletal Pain; Pain | interventions — Acupuncture, Ear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pain Patients
  Interventions: Device: Ear acupuncture

INTERVENTIONS:
Device: Ear acupuncture — Ear acupuncture

SUMMARY:
The purpose of this study is twofold: 1) to test the feasibility of integrating a simple bilateral ear acupuncture procedure (Auricular Stimulation Procedure - ASP) into the standard care delivered in the Aeromedical Evacuation system and 2) to observe and document any changes in pain scores and in-flight related symptoms and factors (e.g. sinus block/pain, ear block pain, nausea/air sickness) typically monitored during transportation of wounded warriors from Ramstein Air Base (RAB) to Andrews Air Force Base (AAFB).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* NRS Pain rating > 0
* Military beneficiaries undergoing aeromedical evacuation from RAB to AAFB

Exclusion Criteria:

* Medically unstable or otherwise unable to participate including those with the inability to consent
* Allergy to metals
* Ear trauma
* Sepsis
* Unhealed wounds on the ears
* Piercing or scar tissue in any of the ear acupuncture point areas
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Military beneficiaries undergoing aeromedical evacuation from Ramstein Air Base to Andrews Air Force Base who are experiencing pain.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Pain | March 2013

CONTACTS AND LOCATIONS:
Overall Officials: Richard Niemtzow, MD, PhD, MPH, Principal Investigator — United States Air Force
Locations (1):
- Ramstein Air Base, Ramstein, Germany